CLINICAL TRIAL: NCT02952027
Title: Evaluating the Effectiveness of Incentive Spirometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Adam Eltorai, Research Fellow, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Lifespan
Record Dates: First submitted 2016-10-18; First posted 2016-11-02 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Dyspnea; Respiratory Rate; Oxygen Saturation; Oxygen Requirements; FEV1; FVC; Atelectasis; Pneumonia; Re-intubation; Hospital Length of Stay; Nursing Workload; Incentive Spirometry
MeSH Terms: conditions — Dyspnea; Pulmonary Atelectasis; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Bell On (Experimental): Subjects in the Bell On arm will receive a timer where the alarm will sound every hour.
  Interventions: Behavioral: Use-recording, patient-reminder alarm for incentive spirometry
- Bell Off (Placebo Comparator): Subjects in the Bell Off arm will receive a timer where the alarm will not sound, but still record incentive spirometer usage
  Interventions: Behavioral: Use-recording, patient-reminder alarm for incentive spirometry

INTERVENTIONS:
Behavioral: Use-recording, patient-reminder alarm for incentive spirometry

SUMMARY:
Post-operative pulmonary complications (PPCs) have a major impact on patients and healthcare expenses. The goal of perioperative respiratory therapy is to improve airway clearance, increase lung volume, and mitigate atelectasis. Incentive spirometers (IS) are ubiquitously used to prevent atelectasis and PPCs-implementation of which requires substantial provider time and healthcare expenses. However, meta-analyses have demonstrated that the effectiveness of ISs is unclear due to poor patient compliance in past studies.

The goal of this investigation is evaluate the effectiveness of IS on post-operative clinical outcomes. The aims of this investigation are to evaluate 1) if IS use compliance can be improved by adding a use-recording patient reminder alarm, and 2) the clinical outcomes of the more compliant IS users vs. the less-compliant IS users.

ELIGIBILITY:
Inclusion Criteria:

* Undergoes any cardiothoracic surgery
* Is transferred to the cardiothoracic surgery intermediate (step-down) unit at Rhode Island Hospital
* Already prescribed an incentive spirometer as standard-of-care
* Followed by any healthcare provider
* Ability to sign informed consent and comply with all study procedures including follow-up for up to 1 year

Exclusion Criteria:

* <18 years of age
* Vulnerable population who in the judgment of the investigator is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-08; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Compliance - Does the alarm improve IS use compliance? | up to 1 week postoperatively
  The primary outcome will be to compare subjects' absolute IS usage count and hourly percent compliance in the Bell On arm vs the Bell Off arms.

SECONDARY OUTCOMES:
Outcomes - Does IS use compliance improve clinical outcomes? | up to 1 week postoperatively
  * Subjective American Thoracic Society's Dyspnea Index43 - administered daily in ICTU
    * ICTU Day 1: Baseline Dyspnea Index
    * ICTU Day 2 through discharge: Transition Dyspnea Index
  * Objective Trend during ICTU stay
    * Vital signs (T, HR, RR, BP)
    * O2 saturation
    * Oxygen requirements
    * CBC Bedside Pulmonary Function Tests (Micro 1, Carefusion)
    * Daily FEV1, FVC, FEV6, PEF, FEV1/FVC, FEV1/FEV6 and F25-75 ratios. Wilcox atelectasis severity score44, 45
    * Scored 0-5 by daily chest x-ray
    * Collaboration with Dr. Terrance Healy, Chief of Chest Radiology, RIH Pneumonia
    * Rate of physician-diagnosed pneumonia
    * Pneumonia severity index48 Length of ICTU stay Mortality
    * In-hospital
    * 30 day post-discharge 30-day readmission rates

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Freitas ER, Soares BG, Cardoso JR, Atallah AN. Incentive spirometry for preventing pulmonary complications after coronary artery bypass graft. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD004466. doi: 10.1002/14651858.CD004466.pub3. PMID 22972072
- [Background] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Background] Narayanan AL, Hamid SR, Supriyanto E. Evidence regarding patient compliance with incentive spirometry interventions after cardiac, thoracic and abdominal surgeries: A systematic literature review. Can J Respir Ther. 2016 Winter;52(1):17-26. PMID 26909010
- [Background] Joyce CJ, Baker AB. What is the role of absorption atelectasis in the genesis of perioperative pulmonary collapse? Anaesth Intensive Care. 1995 Dec;23(6):691-6. doi: 10.1177/0310057X9502300606. PMID 8669602
- [Background] Qaseem A, Snow V, Fitterman N, Hornbake ER, Lawrence VA, Smetana GW, Weiss K, Owens DK, Aronson M, Barry P, Casey DE Jr, Cross JT Jr, Fitterman N, Sherif KD, Weiss KB; Clinical Efficacy Assessment Subcommittee of the American College of Physicians. Risk assessment for and strategies to reduce perioperative pulmonary complications for patients undergoing noncardiothoracic surgery: a guideline from the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):575-80. doi: 10.7326/0003-4819-144-8-200604180-00008. PMID 16618955
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Ephgrave KS, Kleiman-Wexler R, Pfaller M, Booth B, Werkmeister L, Young S. Postoperative pneumonia: a prospective study of risk factors and morbidity. Surgery. 1993 Oct;114(4):815-9; discussion 819-21. PMID 8211699
- [Background] Shander A, Fleisher LA, Barie PS, Bigatello LM, Sladen RN, Watson CB. Clinical and economic burden of postoperative pulmonary complications: patient safety summit on definition, risk-reducing interventions, and preventive strategies. Crit Care Med. 2011 Sep;39(9):2163-72. doi: 10.1097/CCM.0b013e31821f0522. PMID 21572323
- [Background] Khan NA, Quan H, Bugar JM, Lemaire JB, Brant R, Ghali WA. Association of postoperative complications with hospital costs and length of stay in a tertiary care center. J Gen Intern Med. 2006 Feb;21(2):177-80. doi: 10.1111/j.1525-1497.2006.00319.x. PMID 16606377
- [Background] Agostini P, Singh S. Incentive spirometry following thoracic surgery: what should we be doing? Physiotherapy. 2009 Jun;95(2):76-82. doi: 10.1016/j.physio.2008.11.003. Epub 2009 Mar 3. PMID 19627688
- [Background] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401
- [Derived] Eltorai AEM, Baird GL, Eltorai AS, Healey TT, Agarwal S, Ventetuolo CE, Martin TJ, Chen J, Kazemi L, Keable CA, Diaz E, Pangborn J, Fox J, Connors K, Sellke FW, Elias JA, Daniels AH. Effect of an Incentive Spirometer Patient Reminder After Coronary Artery Bypass Grafting: A Randomized Clinical Trial. JAMA Surg. 2019 Jul 1;154(7):579-588. doi: 10.1001/jamasurg.2019.0520. PMID 30969332